CLINICAL TRIAL: NCT00437606
Title: A Nonrandomized, Open Label Study to Examine the Effect of Hepatic Impairment on the Pharmacokinetics/Pharmacodynamics and Safety/Tolerability of GK Activator (2) in Patients With Type 2 Diabetes.'
Brief Title: A Study of the Pharmacokinetics/Pharmacodynamics of GK Activator (2) in Type 2 Diabetes Patients With Hepatic Impairment.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Clinical Trials, Study Director, Hoffmann-La Roche
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP20131
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ethanol

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: GK Activator (2)
- 2 (Experimental)
  Interventions: Drug: Ethanol
- 3 (Experimental)
  Interventions: Drug: GK Activator (2); Drug: Ethanol

INTERVENTIONS:
Drug: GK Activator (2) — 100mg po
  Arms: 1; 3
Drug: Ethanol — 40g po
  Arms: 2; 3

SUMMARY:
This study will investigate the effect of hepatic impairment on the pharmacokinetics, pharmacodynamics, safety and tolerability of GK Activator (2) in type 2 diabetes patients with mild and moderate hepatic impairment. Patients with type 2 diabetes, and with normal hepatic function, or mild or moderate hepatic impairment, will receive a single dose of GK Activator (2) 100mg po before breakfast, for assessment of pharmacokinetic, pharmacodynamic and safety parameters. The anticipated time on study treatment is <3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* type 2 diabetes;
* normal hepatic function, or mild or moderate hepatic impairment.

Exclusion Criteria:

* type 1 diabetes, or latent autoimmune diabetes in adults;
* diabetic neuropathy, retinopathy or nephropathy;
* treatment with insulin or PPAR gamma agonist within 6 weeks of screening;
* clinically significant cardiovascular disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
AUCo-inf and Cmax of plasma and urine GK Activator (2) and M4. AUC0-6 of plasma glucose. | Days 1, 8 and 15

SECONDARY OUTCOMES:
tmax, AUC0-6, AUC0-last, t1/2, CL/F, Ac, CL for GK Activator (2) and M4. Cmin, Cmax, tmax and tmin of plasma glucose. | Days 1, 8 and 15
AEs, laboratory parameters. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Germany (2):
  - Berlin
  - Kiel
- Bratislava, Slovakia